CLINICAL TRIAL: NCT04475978
Title: Intravascular Ultrasound Versus Angiography Guided Drug-coated Balloon Treatment for STEMI Patients：a Prospective, Multicenter, Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020YLK5
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-07

CONDITIONS: STEMI
Keywords: STEMI; drug-coated balloon; IVUS
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVUS group (Experimental)
  Interventions: Device: IVUS-guide DCB PTCA
- Angio group (Placebo Comparator)
  Interventions: Device: Angio-guide DCB PTCA

INTERVENTIONS:
Device: IVUS-guide DCB PTCA — IVUS-guide DCB PTCA
  Arms: IVUS group
Device: Angio-guide DCB PTCA — Angio-guide DCB PTCA
  Arms: Angio group

SUMMARY:
Objectives: The present study aimed to investigate the difference in late luminal loss (LLL) at 9-month after drug-coated balloon (DCB) treatment with intravascular ultrasound (IVUS) versus angiography for ST-segment elevated myocardial infarction （STEMI）patients.

Background: In primary percutaneous coronary intervention for STEMI, DCB angioplasty has proved to be a safe and feasible strategy. Compare with angiography guidance, IVUS-guided PCI significantly improve clinical outcome. With IVUS guidance, STEMI patients undergo DCB angioplasty might have be beneficial results.

Methods: A total of 208 STEMI patients who required DCB treatment were randomly assigned either an IVUS guidance and angiography guidance group. The primary endpoint was late luminal loss at 9-month. Stent thrombosis (ST) was the safety endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction eligible for PPCI:

  1. >20 min of chest-pain and at least 1 mm ST-elevation in at least two contiguous leads, a new left bundle branch block or a true posterior myocardial infarction (confirmed by ECG or echocardiography) .
  2. Reperfusion is expected to be feasible within 12 h after onset of complaints.
* Infarct related artery eligible for PPCI and:

  1. De novo lesion in a native coronary artery
  2. Reference-vessel diameter 2.5 mm and 4 mm
  3. Diameter stenosis of >50% (by visual assessment) after thrombus aspiration and pre-dilatation.

Exclusion Criteria:

* - Age <18 yr and >85 yr
* History of myocardial infarction
* lesion length > 30m
* Left Main lesion
* Ostial lesion
* None-target vessel need to treat with PCI
* Severe calcification
* Severe tortuosity
* Severe angulation
* Cardiogenic shock before pre-dilation or any serious cases can not perform IVUS
* Known contraindication/resistance for bivalirudin, fondaparinux, heparin, aspirin, prasugrel and/or ticagrelor
* Participation in another clinical study, interfering with this protocol Uncertain
* Known intracranial disease (mass, aneurysm, AVM, haemorrhagic CVA, ischemic CVA/TIA <6 months before inclusion or ischemic CVA with permanent neurological deficit) Gastrointestinal/urinary tract
* bleeding <2 months before inclusion Refusal to receive blood transfusion
* Planned major surgery within 6 weeks
* Stent implantation <1 week before inclusion
* Expected mortality from any cause within the next 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
late lumen loss（LLL） | At 9 months follow-up
  late lumen loss（LLL）

SECONDARY OUTCOMES:
target lesion failure (TLF) | At 1-year follow-up
  the composite of car- diac death, target-vessel MI (TVMI), or clinically driven TLR

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Zhou, Ph.D, Principal Investigator — Clinical Trial Center of Xiamen Cardiovascular Hospital
Locations (1):
- Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian, China